CLINICAL TRIAL: NCT01114087
Title: Impact of the Inhibitors of Tyrosine Kinase on the Male Fertility
Acronym: GLIFERTI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Amel Ouslimani, Department Clinical Reseach of Developpement
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P070131
Record Dates: First submitted 2010-04-29; First posted 2010-04-30 (Estimated); Last update posted 2011-03-29 (Estimated); Status verified 2011-01

CONDITIONS: Chronic Myeloid Leukemia; Gastrointestinal Stromal Tumors
Keywords: Spermatogenesis; Inhibitors of tyrosine kinase; Fragmentation of the spermatic DNA
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Gastrointestinal Stromal Tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Patients presenting with chronic myeloid leukaemia or malignant GIST and receiving for the first time a treatment by imatinib, a tyrosin-kinase inhibitor, preceded or not by hydroxyurea therapy for less than one month.
  Interventions: Drug: Imatinib treatment

INTERVENTIONS:
Drug: Imatinib treatment — Imatinib is a tyrosin-kinase inhibitor

SUMMARY:
Evaluate the possible deleterious effects of tyrosine kinase inhibitors on sperm concentration, after 6 months of therapy, which corresponds to 2 cycles of spermatogenesis and on the sperm nuclear integrity. The main comparison criterion will be the mean difference in sperm concentration before and after the 6 month treatment.

DETAILED DESCRIPTION:
Antityrosine - kinases, such as imatinib are presently the gold standard therapy of chronic myeloid leukaemia (CML), with complete cytogenetic responses being achieved in 70-90% of patients receiving the drug as first -line monotherapy. Imatinib selectively inhibits the hybrid oncogen BCR/ABL involved in the genesis of CML and other tyrosine kinases, such as c-kit and platelet derived growth factor receptor (PGDF-R), involved in malignant gastro intestinal stromal tumours (GIST) . Despite its good tolerance, in vivo animal studies have proved that imatinib induces teratogenesis and dose-related effect on spermatogenesis. In humans, few pregnancies involving male CML patients have been reported with one spontaneous abortion, one case of gut malrotation and 15 healthy children. However, in the absence of detailed and definite evidence of the lack of deleterious effect of imatinib on spermatogenesis and sperm nuclear integrity in humans, specific studies are warranted. Male patients (38) will be included in this study if they are 18 to 60 years old, presenting with chronic myeloid leukaemia or malignant GIST and receiving for the first time a treatment by imatinib, a tyrosin-kinase inhibitor, preceded or not by hydroxyurea therapy for less than one month. These patients should have signed the informed consent and be covered by the French social security system. In this open prospective study, each patient will be his own control. The effect of imatinib on the spermatogenesis will be evaluated by the concentration of spermatozoa before the beginning of the treatment and after 6 months of imatinib, representing 2 cycles of spermatogenesis. Patients will be recruited by the onco-haematologists (5 corresponding centres) and referred to the CECOS Tenon. A medical investigator will collect the informed consent and fill the study file. A classical sperm analysis, according to OMS, will be performed. A sample of the ejaculate will be fixed for further analysis of the percentage of sperm nuclei with fragmented DNA (TUNEL procedure). The rest of the semen will be frozen, packaged in straws and stored in liquid nitrogen to be used, if necessary, by the patient if an ART is mandatory to conceive a child.Another sperm recovery will be performed after a period of 6 months under the anti tyrosine-kinase (ATK) therapy and the same sperm analysis will be carried out and the results compared to the first evaluation, before ATK. The plasmatic concentration of imatinib will be determined, for each patient, the day of the second sperm recovery to check the efficiency of ATK administration.

ELIGIBILITY:
Inclusion Criteria:

* Men from 18 to 60 years old
* Patients recently diagnosed CML or GIST
* Patients for whom a treatment by an inhibitor of tyrosine kinase in monotherapy is prescribed
* Patients having signed the informed consent
* Patients with social security

Exclusion Criteria:

* Patients already subjected to a treatment potentially sterilizing
* Patients under supervision or guardianship

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 2 (Actual)
Dates: Start 2008-10; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Average difference of the concentration of spermatozoa in the ejaculate measured before treatment and after 6 months of treatment. | At the inclusion and M6 visits

SECONDARY OUTCOMES:
Analysis of the fragmentation of the spermatic DNA | At the inclusion and M6 visits
Plasmatic concentration of the inhibitors of tyrosine kinase | At the inclusion and M6 visits

CONTACTS AND LOCATIONS:
Overall Officials: Jacqueline Mandelbaum, Dr, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- Department of Biology of reproduction (TENON Hospital-APHP), Paris, France